CLINICAL TRIAL: NCT02924909
Title: Phase II Trial of Induction Chemotherapy Followed by Chemoradiotherapy With Paclitaxel and Carboplatin Before Minimal Invasive Surgery in Patients With Localized Esophageal and Gastro-esophageal Junction Cancer
Brief Title: Phase II Trial of Neoadjuvant Treatment and Minimal Invasive Surgery for Esophageal and GEJ Cancer
Acronym: QUIMERA
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto Nacional de Cancer, Brazil (Other Government)
Responsible Party: Principal Investigator, Mariana Bruno Siqueira, Principal Investigator, Instituto Nacional de Cancer, Brazil
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 54633416.3.0000.5274
Record Dates: First submitted 2016-08-31; First posted 2016-10-05 (Estimated); Last update posted 2018-03-20 (Actual); Status verified 2018-03

CONDITIONS: Esophageal Cancer; Induction Chemotherapy
MeSH Terms: conditions — Esophageal Neoplasms | interventions — CP protocol; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- induction carboplatin paclitaxel (Experimental): carboplatin AUC=6 21 day cycle for 2 cycles paclitaxel 175 mg/m2 21 day cycle for 2 cycles radiotherapy 4500 cGy in 25 fractions carboplatin AUC=2 in a week regimen during radiotherapy paclitaxel 50 mg/m2 in a week regimen during radiotherapy Minimal Invasive Surgery
  Interventions: Drug: carboplatin paclitaxel

INTERVENTIONS:
Drug: carboplatin paclitaxel — induction carboplatin paclitaxel for 2 cycles
  Other Names: Taxol, Carbo

SUMMARY:
Phase II trial of induction chemotherapy with carboplatin AUC 6 plus paclitaxel 175 mg/m2 in a 21 day cycle for two cycles followed by radiotherapy 4500 cGy in 25 fractions plus carboplatin AUC=2 paclitaxel 50 mg/m2 in a week regimen followed by minimally invasive surgery after 6 to 10 weeks. A PET scan will be performed at the time of randomization and 14 days after de first cycle to determine the relation between metabolic response and survival.

DETAILED DESCRIPTION:
Phase II trial of induction chemotherapy with carboplatin AUC 6 plus paclitaxel 175 mg/m2 in a 21 day cycle for two cycles followed by radiotherapy 4500 cGy in 25 fractions plus carboplatin AUC=2 paclitaxel 50 mg/m2 in a week regimen followed by minimally invasive surgery after 6 to 10 weeks. A PET scan will be performed at the time of randomization and 14 days after de first cycle to determine the relation between metabolic response and survival. The primary endpoint is to the evaluate the number of complete pathologic response. The secondary endpoints are evaluation of toxicity, radiologic response, metabolic response, results of the minimally invasive surgery (blood lost, number of conversion to open surgery, type of resection, R0, 1 or 2, post-op complications, time of hospitalization, 30 day post-op mortality), evaluate the viability of treatment protocol (number of patient that complete the phases), evaluate quality of life during the treatment and after the surgery. Inclusion criterias are: Histologically proven adenocarcinoma or squamous cell carcinoma of the middle and lower third of the esophagus (included tumors located in the gastro-esophageal junction Siewert I and II), age between 18 and 75 years, Performance Status 0 or 1, neutrophils count > 1500/mm3, platelets count > 100.000/mm3, hemoglobin count > 9 g/dL, preserve hepatic and renal function, stage (TNM AJCC 7th edition): cT1b-3, N0-1, M0, signature of the informed consent. Exclusion criterias are: history of another cancer, except skin non melanoma, pregnancy or history of hypersensitivity to the study drugs

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven adenocarcinoma or squamous cell carcinoma of the middle and lower third of the esophagus (included tumors located in the gastro-esophageal junction Siewert I and II)
* Age between 18 and 75 years
* Performance Status 0 or 1
* Stage (TNM AJCC 7th edition): cT1b-3, N0-1, M0

Exclusion Criteria:

* History of another cancer, except skin non melanoma
* Pregnancy
* History of hypersensitivity to the study drugs

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-02-01 (Actual); Primary Completion 2020-09 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
complete pathological response | 2 weeks after surgery
  complete pathological response will be evaluate in the surgical specimen after the neoadjuvant treatment

CONTACTS AND LOCATIONS:
Overall Officials: Mariana Siqueira, MD, Principal Investigator — INCA Brazil
Locations (1):
- INCA- Instituto Nacional de Câncer, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No